CLINICAL TRIAL: NCT01015560
Title: S0916, A Phase II, Window Trial of the Anti-CCR2 Antibody MLN1202 in Patients With Bone Metastases
Brief Title: S0916, MLN1202 in Treating Patients With Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0916; S0916 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: bone metastases; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis | interventions — plozalizumab; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): MLN1202 8mg/kg IV Days 1, 15, 29 given as 1 6 week cycle
  Interventions: Drug: anti-CCR2 monoclonal antibody MLN1202; Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: anti-CCR2 monoclonal antibody MLN1202
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such MLN1202, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well MLN1202 works in treating patients with bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the urinary n-telopeptide (uNTX) response to anti-CCR2 monoclonal antibody MLN1202 in patients with bone metastases.

Secondary

* To assess the feasibility of performing cross-disease site trials within the Southwest Oncology Group.
* To explore the effect of anti-CCR2 monoclonal antibody MLN1202 on markers of tumor cell proliferation, monocytes/macrophage trafficking, and osteoclast maturation.
* To estimate allele frequencies of defined SNPs occurring in the CCL2 and CCR2 genes in these patients.

OUTLINE: This is a multicenter study.

Patients receive anti-CCR2 monoclonal antibody MLN1202 IV over 1 hour on days 1, 15, and 29 in the absence of disease progression or unacceptable toxicity.

Patients undergo urine and blood sample collection at baseline and on days 15, 29, and 43 for correlative biomarker and polymorphism studies.

After completion of study treatment, patients are followed up for ≥ 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiographically documented metastases to the bone by bone scan, x-ray, CT scan, MRI, or PET scan within the past 42 days

  * Documentation of progression of metastatic disease by serial scans is not required for study entry
* No untreated or progressive brain metastases

  * History of brain metastases allowed provided they have been treated and remain controlled

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must consent to urine and blood specimen submissions
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with the study requirements
* No known hypersensitivity to anti-CCR2 monoclonal antibody MLN1202 or other recombinant human antibodies

PRIOR CONCURRENT THERAPY:

* At least 14 days since prior radiotherapy and recovered (≤ grade 1 from all related toxicities)
* At least 84 days since prior radionuclide therapy (e.g., strontium, samarium) and recovered (≤ grade 1 from all related toxicities)
* More than 14 days since prior investigational agents, chemotherapeutic agents, or other anticancer agents
* Concurrent bisphosphonate therapy for bone metastases allowed provided treatment was initiated ≥ 28 days before study entry

  * No initiation of bisphosphonates during study treatment
* Concurrent hormonal therapy (e.g., anti-estrogens or anti-androgens) or stable doses of steroids for cancer allowed provided treatment was initiated > 14 days before study entry
* No concurrent G-CSF or other growth factor support

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Pienta, MD, FACP, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (47):
- United States (47):
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- MLN 1202: MLN1202 8mg/kg IV Days 1, 15, 29 given as one 6-week cycle
Period: Overall Study
Arm/Group | MLN 1202
Started | 44
Eligible and Analyzable | 43
Completed | 41
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Not protocol specified | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Eligible and analyzable patients included.
Arm/Group | MLN 1202
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39
  Black | 4

OUTCOME MEASURES:

1. Primary Outcome: uNTX Response Rate at 43 Days
Description: Urinary n-telopeptide (uNTX) response is defined as a 25% reduction from baseline levels. Patients with missing response data were included as non-responders.
Time Frame: 43 days
Population: Eligible and analyzable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MLN 1202
Number analyzed (Participants) | 43
percentage of participants | 14 [5 to 27]

ADVERSE EVENTS:
Time Frame: Minimum of 30 days after the last dose of protocol therapy, or every 4 to 6 weeks until all protocol therapy-related toxicities resolve, return to baseline, or are deemed irreversible, whichever is longer.
Description: Only eligible and analyzable patients that were assessed for adverse events are included. One patient was not assessed for adverse events and is not included in this analysis.
Arm/Group | MLN 1202
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 30/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN 1202 (N=42)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN 1202 (N=42)
Anemia (Blood and lymphatic system disorders) | 10
Diarrhea (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 15
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
CD4 lymphocytes decreased (Investigations) | 4
Creatinine increased (Investigations) | 8
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Urinary frequency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No